CLINICAL TRIAL: NCT02880137
Title: (RTMPE for CAV) Real Time Myocardial Perfusion Echocardiography for Detection of Coronary Allograft Vasculopathy in Cardiac Transplant Patients
Brief Title: Real Time Myocardial Perfusion Echocardiography for Coronary Allograft Vasculopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Jonathan N. Johnson, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-007825
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Allograft Vasculopathy
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RTMPE (Experimental): RTMPE with Perflutren Lipid Microsphere (DEFINITY) is a safe and feasible non-invasive technique commonly used to diagnose coronary disease, and offers an attractive alternative for CAV detection.
  Interventions: Drug: Perflutren Lipid Microsphere; Procedure: RTMPE

INTERVENTIONS:
Drug: Perflutren Lipid Microsphere — Definity (injectible suspension ultrasound contrast agent) will be diluted with saline for both Pediatric and Adult subjects. For pediatric subjects under 60kg (kilogram), the dose will be 20 MicroL/kg (MicroLiter/kilogram) diluted to the same concentration used in the adult dosing. Hand Injections will be performed at baseline, Pre-peak, and peak perfusion stages.
  Other Names: Definity
Procedure: RTMPE — Utilizes intravenous administration of biologically-inert microbubbles to assess myocardial perfusion and has demonstrated utility for identifying small vessel coronary artery disease.
  Other Names: Real Time Myocardial Perfusion Echocardiography

SUMMARY:
Is real-time myocardial perfusion echocardiography (RTMPE) a feasible and effective non-invasive method to detect significant Coronary Allograft Vasculopathy in pediatric and adult cardiac transplant recipients? Will perfusion deficits correlate with significant coronary artery stenosis identified by standard stress echocardiography and Invasive Coronary Angiography (ICA), and identify diffuse small vessel disease more effectively than current non-invasive techniques?

DETAILED DESCRIPTION:
Heart transplant recipients are susceptible to developing a unique disease that causes blockages in the arteries of the transplanted heart (coronary arteries) called Coronary Allograft Vasculopathy (CAV). Because CAV often progresses without symptoms, transplant recipients undergo regular surveillance testing so that CAV can be detected and treatment can be offered before significant damage to the transplanted heart occurs. Current tests used to detect CAV are either invasive (with risk of complications) or may not be able to detect CAV in its early stages. Myocardial contrast perfusion echocardiography is a safe non-invasive diagnostic test that may be well suited for detecting CAV, however has not been well studied in heart transplant recipients. This study examines the ability of myocardial contrast perfusion echocardiography to detect CAV in adult and pediatric heart transplant recipients, and compare those results to current standard testing strategies such as Invasive Coronary Angiography (ICA) and standard stress echocardiography. This will help determine whether myocardial contrast perfusion echocardiography is a better test for regular surveillance of CAV in adult and pediatric transplant recipients.

ELIGIBILITY:
Inclusion:

* Cardiac transplant recipients (> or equal to 10 months post transplant)
* Clinically followed at Mayo Clinic, Rochester Minnesota

Exclusion:

* Standard contraindications to the use of ultrasound contrast and pharmacologic stress
* Recent (< 3 months) hospitalization for heart failure, acute coronary syndrome or allograft rejection
* Multi-organ transplant Known or suspected right-to-left, bi-directional, or transient right-to-left cardiac shunts
* Hypersensitivity to perflutren

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan N Johnson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Nowell Fine University of Calgary 1403 29th Street NW Canada
  Researchers at University of Calgary are also conducting this study and will collaborate with Mayo Clinic on the research data.
  Study identification number, subject Identification, or any other unique identifying number, characteristic, or code that the external party is unable to link to the identity of the subject. Dates: all elements of dates [month, day, and year] directly related to an individual, e.g. date of birth, death, or diagnosis, etc. City, county, precinct, zip code, and their equivalent geocodes.

RESULTS

PARTICIPANT FLOW:
Groups:
- RTMPE: RTMPE with Perflutren Lipid Microsphere (DEFINITY) is a safe and feasible non-invasive technique commonly used to diagnose coronary disease, and offers an attractive alternative for cardiac allograft vasculopathy (CAV) detection.
  Perflutren Lipid Microsphere: Definity (injectible suspension ultrasound contrast agent) will be diluted with saline for both Pediatric and Adult subjects. For pediatric subjects under 60kg (kilogram), the dose will be 20 MicroL/kg (MicroLiter/kilogram) diluted to the same concentration used in the adult dosing. Hand Injections will be performed at baseline, Pre-peak, and peak perfusion stages.
  RTMPE: Utilizes intravenous administration of biologically-inert microbubbles to assess myocardial perfusion and has demonstrated utility for identifying small vessel coronary artery disease.
Period: Overall Study
Arm/Group | RTMPE
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RTMPE
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27
  Canada | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Perfusion Defect
Description: A perfusion defect will first be identified using clinically indicated invasive coronary angiography (ICA). The presence of a perfusion defect will then be identified using non-invasive real time myocardial perfusion echocardiography (RTMPE).
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | RTMPE
Number analyzed (Participants) | 36
Participants
  Perfusion defect identified by ICA | 5
  Perfusion defect identified by RTMPE | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the duration of the echocardiogram, approximately 40 minutes.
Arm/Group | RTMPE
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT02880137/Prot_SAP_000.pdf